CLINICAL TRIAL: NCT07128277
Title: Clinical Study of Trap (FAPI) 3 PET Imaging in Noninvasive Diagnosis of Malignant Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xiao Chen, Director of Nuclear Medicine Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 2025179
Record Dates: First submitted 2025-08-13; First posted 2025-08-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — histopathological findings obtained from biopsy or resected surgical specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with malignant tumors: a) Age between 18 and 65 years, gender not limited; b) Patients with malignant tumors confirmed by biopsy or surgical pathology; c) Imaging findings of suspicious lymph nodes or distant metastases; d) Written informed consent from the subject or his/her legal guardian.

SUMMARY:
Positron Emission Tomography (PET) is a functional imaging technology for diagnosing and monitoring tumors. In clinical applications for malignant tumors, PET includes staging, response assessment, and prognosis prediction, providing attractive semi-quantitative biomarkers for both clinical and research platforms. Understanding the fundamentals of imaging science and evaluating the strengths and limitations of imaging modalities is crucial for optimizing research assessments. With the widespread use of functional techniques and the development of novel PET biomarkers, PET-based research evaluations will be further enhanced. The field of oncology has undergone a revolution through molecular imaging, which evaluates tumor biology, while traditional radiological imaging focuses on morphological anatomy . Molecular imaging employs non-invasive visualization at cellular or subcellular levels to observe physiological or pathological processes, whereas PET/CT serves as a hybrid imaging tool that provides complementary information on both function and structure . [18F] Fluorodeoxyglucose (FDG), first developed in the late 1970s as a tracer for brain region metabolism, remains the most widely used PET tracer with diverse applications in both oncology and non-oncology fields . Despite its undeniable clinical utility, FDG uptake serves as an alternative indicator for glucose transport/metabolism rather than being specific to malignant tumors. Continuous exploration of cellular targets has led to the discovery of fibroblast activation protein (FAP). Cancer-associated fibroblasts are present in many tumors, particularly those with strong fibrotic-promoting responses such as breast cancer, colorectal cancer, pancreatic cancer, prostate cancer, and lung cancer. Consequently, FAP expression has been observed in over 90% of epithelial tumors. To date, FAP expression has been associated with poor tumor prognosis in colorectal cancer, pancreatic cancer, hepatocellular carcinoma, and ovarian cancer . Although more research is needed, this advantage makes cancer-associated fibroblasts an ideal target for anti-tumor therapy. In practical applications, low FAP expression in fibroblasts or healthy tissues facilitates imaging of subtle pathological changes. Cancer-associated fibroblasts (CAFs), a key component of the tumor microenvironment, account for over half the mass in various tumor types. Previous studies indicate that CAFs play significant roles in tumor growth, immune suppression, and cancer invasion . Therefore, CAFs may become emerging targets for tumor diagnosis and treatment. Fibroblast activation protein (FAP) is overexpressed in CAFs of multiple epithelial cancers but shows weak expression in healthy tissues, making it a promising target in cancer research. Recent years have seen expanded molecular imaging studies targeting FAP in tumor diagnosis . The excellent tumor-targeting efficacy of FAP has been confirmed through multiple clinical trials . The results clearly establish FAPI as a highly promising tumor-targeting ligand with significant potential applications in translational oncology. However, its therapeutic efficacy remains under investigation. An ideal radiopharmaceutical for cancer treatment should demonstrate excellent targeting specificity and relatively long tumor retention time. Previous studies have shown that radiolabeled FAPI variants (FAPI-04 and FAPI-46) accumulate rapidly and satisfactorily in tumors while showing low physiological uptake in normal tissues. However, previous FAP-related tracers exhibited relatively short tumor retention times . Our aim is to design a FAPI trimer, Trap-(FAPI)3, to optimize pharmacokinetics and evaluate whether this novel drug demonstrates superior advantages over its monomeric analogs in tumor imaging diagnosis and staging.

DETAILED DESCRIPTION:
4.1 Research Site and Population This study enrolled patients with confirmed malignant tumors at the Army Specialized Medical Center between April 2025 and April 2027, as verified by biopsy or surgical pathology. 4.2 Sample Size Determination Using PASS software, the investigators calculated the required sample size by selecting the "Test for a single-sample Sensitivity and Specificity" under Diagnostic Tests (ROC). Based on prior literature and pilot studies, the sensitivity (Sensitivity) of 18F RCCB6 imaging for predicting treatment efficacy was estimated at 85%, with a specificity (Specificity) of 75%. With confidence levels α=0.05, β=0.2, and p=0.25, the null hypotheses for both sensitivity and specificity were set at 50%. Data analysis yielded a required sample size of 32.4.3 Survey Content 4.3.1 Clinical Data Collection All patients' disease progression, laboratory tests (tumor markers), pathological findings, and relevant immunohistochemical data were recorded. Image analysis and observation metrics: Trap- (FAPI) 3 PET/CT or PET/MR images were independently reviewed and processed by two experienced nuclear medicine physicians. The following indicators were recorded and evaluated: 1) Visual image analysis: including lesion location, size, morphology, and uptake extent; 2) Semi-quantitative analysis: measuring standard uptake value (SUV) of lesions and the ratio between lesion SUV and liver/blood pool SUV. 4.3.3 Pathological Analysis After collecting pathological specimens from primary lesions and metastatic lymph nodes post-surgery, formalin fixation and paraffin embedding were performed before sectioning into 4μm-thick slices for FAP staining. 4.4 Data Management and Statistical Analysis The Department of Nuclear Medicine at the Army Specialized Medical Center was responsible for data management and analysis. A spreadsheet system was established to centrally manage all enrolled patients 'basic information, laboratory tests, PET/CT/MR imaging results, postoperative pathology, and immunohistochemistry. Original PET/CT/MR images of all enrolled patients were archived. Statistical analysis was conducted using SPSS20.0 software. Qualitative data were presented as frequency using chi-square or Fisher's exact test. Quantitative data were analyzed using Kolmogorov-Smirnov normality tests, with normally distributed data expressed as (x±s). Independent samples t-tests were employed for normal distribution verification; non-normal distribution data were represented by median (upper/lower quartiles) using Wilcoxon rank sum tests. Pearson correlation analysis evaluated the correlation between lesion FAP expression levels and PET imaging. Receiver-operated characteristic (ROC) curves were used to assess diagnostic performance, calculating area under the curve (AUC), sensitivity, specificity, and thresholds for each variable. The diagnostic efficacy of PET/MRI and PET/CT was compared by Medcalc software. P <0.05 was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old, gender is not limited
* Patients with malignant tumors confirmed by biopsy or surgical pathology
* Suspected lymph node or distant metastasis found by imaging
* Written informed consent signed by the subject or his/her legal guardian

Exclusion Criteria:

* Patients receiving anti-tumor therapy prior to PET/CT or PET/MR scans
* Patients with severe medical conditions unable to tolerate PET/CT or PET/MR scans
* Eligible participants with contraindications for PET/CT or PET/MR scans
* Participants with radiation exposure exceeding 50 mSv in the past year
* Participants who underwent major surgery within the last three months or received experimental drugs/instruments (with unclear efficacy/safety) within one month
* Participants with clinical conditions that the study sponsor considers potentially hazardous or harmful to this investigational agent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects we selected are adults who are not restricted by gender. For details, please refer to the "EligibilityCriteria" colymn.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-08-13 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | Completed within half year after end of the study
  The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FDG and 68Ga-Trap-FAPI PET were calculated and compared to evaluate the diagnostic efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan Y, Li J, Zhao T, Zhou M, Liu K, Xiang S, Tang Y, Jakobsson V, Xu P, Chen X, Zhang J. Clinical translation of a novel FAPI dimer [68Ga]Ga-LNC1013. Eur J Nucl Med Mol Imaging. 2024 Jul;51(9):2761-2773. doi: 10.1007/s00259-024-06703-z. Epub 2024 Apr 2. PMID 38561515